CLINICAL TRIAL: NCT03035227
Title: Catheter Ablation of Arrhythmias to Improve CRT Response
Acronym: ABLATE-CRT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left Institution.
Sponsor: Kansas City Heart Rhythm Institute (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003861
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2020-04

CONDITIONS: Arrhythmia, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Catheter Ablation; Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter Ablation (Active Comparator): Catheter ablation procedure of atrial and/or ventricular arrhythmias.
  Interventions: Procedure: Catheter Ablation
- Medical Therapy (Active Comparator): Medical management using antiarrhythmic drugs per standard of care of treating physician.
  Interventions: Drug: Anti-Arrhythmics

INTERVENTIONS:
Procedure: Catheter Ablation — Catheter ablation of atrial or ventricular arrhythmia. The technique and type of ablation will be at the discretion of the treating electrophysiologists.
  Arms: Catheter Ablation
Drug: Anti-Arrhythmics — Anti-Arrhythmic drugs that are deemed to be appropriate for the given participants's arrhythmia by the treating physician.
  Arms: Medical Therapy

SUMMARY:
The purpose of this study is to test if catheter ablation is better than medication therapy at treating arrhythmias originating from the upper and/or lower chambers of the heart in order to allow the heart to beat properly.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients with CRT-D or CRT-P greater than 3 months
* Bi-ventricular pacing less than 94% of the time
* 3 months after CRT-D or CRT-P implantation an EF improvement less than 5%
* Presence of one of the following arrhythmias and eligible for catheter ablation:
* Atrial fibrillation
* Atrial flutter
* Supraventricular tachycardia
* Premature ventricular contraction burden greater than 30% in a 24-hour period
* Ventricular tachycardia

Exclusion Criteria:

* Estimated survival less than one year
* Patient unable to make scheduled follow up visits at treating center
* Participating in another investigational study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Therapy: The medical treatment arm consist of the use of antiarrhythmic drugs that are deemed to be appropriate for the given arrhythmia by the treating physician.
- Ablation Arm: Patients enrolled into the ablation arm will under go catheter ablation of atrial or ventricular arrhythmia within 3 months of signing the informed consent form.
Period: Overall Study
Arm/Group | Medical Therapy | Ablation Arm
Started | 1 | 1
Completed | 0 (study stopped due to PI leaving institution) | 0 (study stopped due to PI leaving institution)
Not Completed | 1 | 1
Not completed — study stopped due to PI leaving institut | 1 | 1

BASELINE CHARACTERISTICS:
Population: data not collected to be analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Catheter Ablation | Medical Therapy | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Change in Ejection Fraction (EF)
Description: Change in Ejection Fraction (EF)
Time Frame: 90 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Bi-ventricular Pacing Improvement
Description: data not analyzed
Time Frame: 90 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Cardiovascular Mortality
Description: data not analyzed
Time Frame: 365Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: All-cause Mortality
Description: data was not analyzed
Time Frame: 365 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hospital Admissions for Heart Failure Exacerbation
Description: data not analyzed
Time Frame: 365 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: New York Heart Association (NYHA) Class Change
Time Frame: 30 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in 6 Minute Walk Test
Description: data not analyzed
Time Frame: 30 Days
Population: data not analyzed
Arm/Group | Medical Therapy | Ablation Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Quality of Life - SF-36
Description: data not analyzed
Time Frame: 30 Days
Population: data not analyzed
Arm/Group | Ablation Arm | Medical Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Quality of Life Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: data not analyzed
Time Frame: 30 Days
Population: data not analyzed
Arm/Group | Ablation Arm | Medical Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed.
Description: Adverse Events were not monitored/assessed. No data collected - enrolled two patients and that is all. Study was cancelled.
Arm/Group | Medical Therapy | Ablation Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT03035227/Prot_SAP_001.pdf